CLINICAL TRIAL: NCT07218484
Title: Feasibility of VoiceLove Digital Therapy for Delirium Management in ICU Patients: A Pilot Study
Brief Title: VoiceLove Digital Therapy for Delirium in the ICU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PRO00041572
Record Dates: First submitted 2025-08-28; First posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Delirium
Keywords: delirium; intensive care unit; cognitive dysfunction; confusion
MeSH Terms: conditions — Delirium; Cognitive Dysfunction; Confusion

STUDY DESIGN:
Intervention Model Description: The study is a single-center, single-arm, prospective trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient participant (Experimental): Two sessions per day of VoiceLove digital therapy will be administered with each session lasting 20-25 minutes. Sessions will occur during days 1-3 while the participant is in bed and in an alert and calm state.
  Interventions: Behavioral: VoiceLove therapy

INTERVENTIONS:
Behavioral: VoiceLove therapy — VoiceLove digital interventions represent voice recordings, specifically, (i) Reorientation messages, and (ii) general communication domain calming and encouraging voice messages recorded in familiar voices from family and friends. Families will be guided to record and deliver Reorientation messages, that can be played to the patient.

SUMMARY:
The study is a single-center, single-arm, prospective trial to evaluate the feasibility, safety, and acceptability of VoiceLOVE digital therapy for the management of delirium in surgical ICU patients. 15 participants will be enrolled. The study expects that 70% of participants will complete 20 -25 minutes of the VoiceLOVE digital therapy. Descriptive statistics will be used to summarize the findings. The intent is that this study will provide information for a larger, subsequent clinical trial of surgical ICU patients who are at risk for delirium.

DETAILED DESCRIPTION:
VoiceLove digital therapy includes voice recordings of the participant's loved one delivered at the bedside via a smartphone attached to the bed. The VoiceLove digital therapy will be delivered in the morning and in the evening and will play for 20-25 minutes each session.

Participants will have a pre-operative visit, 3 consecutive intervention visits with vital signs assessment, 7 days of assessments of Confusion Assessment Methods (CAM)-ICU (morning and evening), and 7 days of a Richmond Agitation-Sedation Scale assessment. The participant will provide an assessment of the acceptability of the VoiceLove digital therapy using a system usability scale score at the end of their participation in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged ≥18 years admitted to the hospital after major surgery (elective or non-elective) require a hospital stay of at least five days following surgery, including an ICU stay for at least three days after the surgical procedure
2. At risk of delirium, as per ICU delirium risk score or existing diagnosis
3. Family members or caregivers involved in patient care at least 18 years of age.
4. Clinical team members caring for the patients

Exclusion Criteria:

* Patients in the ICU who have

  1. a history of severe mental illness,
  2. admission for a drug overdose,
  3. severe vertigo,
  4. a history of severe postoperative nausea and vomiting,
  5. hearing or visual impairments,
  6. preexisting severe dementia (Montreal Cognitive Assessment Score <15),
  7. neurological surgeries.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-08-21 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of VoiceLove digital therapy use by participants in the ICU | Baseline to day 3
  70% of participants complete two 25-minute sessions of VoiceLove digital therapy per day for 3 days

SECONDARY OUTCOMES:
Change in peripheral arterial oxygen saturation (SpO2) after VoiceLove digital therapy | Start of VoiceLove digital therapy to 25 minutes of session on day 1, on day 2, and on day 3.
  Mean change in SpO2 during VoiceLove digital therapy sessions
Change in blood pressure after VoiceLove digital therapy | Start of Voice Love digital therapy to 25 minutes of session on day 1, on day 2, and on day 3.
  Mean change in blood pressure during VoiceLove digital therapy sessions
Change in respiratory rate after VoiceLove digital therapy | Start of VoiceLove digital therapy to 25 minutes of session on day 1, on day 2, and on day 3.
  Mean change in respiratory rate during VoiceLove digital therapy sessions
Change in heart rate after VoiceLove digital therapy | Start of VoiceLove digital therapy to 25 minutes of session on day 1, on day 2, and on day 3.
  Mean change in heart rate during VoiceLove digital therapy sessions

OTHER OUTCOMES:
Acceptability of VoiceLove digital therapy | Day of Hospital Discharge, Visit 8
  Proportion of participants with a system usability scale score >35
Delirium onset during the study | From start of VoiceLove digital therapy sessions at baseline through study completion, day 7
  Proportion of participants with delirium onset
Hypoactive delirium | From start of VoiceLove digital therapy sessions at baseline through study completion, day 7
  Proportion of participants with hypoactive delirium
Hyperactive delirium | From start of VoiceLove digital therapy sessions at baseline through study completion, day 7
  Proportion of participants with hyperactive delirium
Delirium severity | From start of VoiceLove digital therapy sessions at baseline through study completion, day 7
  Proportion of participants with mild, moderate, or severe delirium
Delirium days | From start of VoiceLove digital therapy sessions at baseline through study completion, day 7
  Total number of delirium-positive days
Readmissions to the ICU during the hospital stay | From last day in ICU to a return to ICU prior to hospital discharge, Visit 8
  Total number of readmissions to the ICU
Family satisfaction survey | ICU day 3, Visit 4
  Total score of system usability survey for family or caregiver member

CONTACTS AND LOCATIONS:
Overall Officials: Hina Faisal, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
The study does not allow release of individual participant data